CLINICAL TRIAL: NCT00761176
Title: A Controlled Study Comparing Basic Wound Care to the Provant® Therapy System as an Adjunct to Basic Wound Care for Wound Surface Area Reduction in Diabetic Plantar Foot Wounds
Brief Title: A Pilot Study of the Provant Therapy System in Subjects With Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol Violations noted for 6 of 8 patients
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGI-08-08-1
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetes; Ulcers; Wounds
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Ulcer; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care will be utilized without the device.
- The Provant Therapy System (Other): Thirty minutes, twice daily treatment
  Interventions: Device: The Provant Therapy System

INTERVENTIONS:
Device: The Provant Therapy System — The Provant Wound Therapy System is a safe adjuvant non-invasive medical device.
  Other Names: Radio frequency generator devices
  Arms: The Provant Therapy System

SUMMARY:
The objective of this study is to compare the reduction in wound surface areas between patients with diabetic ulcers utilizing Provant's pulsed radio frequency energy therapy (PRFE) as an adjunct to standardized basic wound care to those utilizing standardized basic wound care alone.

DETAILED DESCRIPTION:
According to the American Diabetes Association (ADA), there are approximately 20.8 million people in the US with diabetes or 7% of the population (1). A significant number of the diabetic population is prone to pedal ulceration and estimates reveal that 15-20% of this population will develop a foot ulcer in their lifetime.

Treatment of diabetic foot ulcerations have posed a problem to healthcare providers for many years. The literature describes many different modalities for direct wound treatment strategies. Most of these treatments rely on the timely application of biological dressings, offloading of the wound, regular (and often inconvenient) visits to the doctor, and most important, compliance by the patient. It is not uncommon for such wounds to be present for greater than six months, despite use of debridement, off-loading and other basic wound care techniques, before presenting for advanced therapy.

Provant has been selected for study because:

* It is already indicated for the adjunctive palliative treatment of postoperative pain and edema in superficial soft tissue.
* It is a non-invasive wound treatment system which utilizes a proprietary PRFE signal which is hypothesized to trigger the release of endogenous growth factors that induce mitosis through accelerating the cell cycle, using a Ca+2 mediated pathway. The result is a significant increase in the rate of cell replication.
* It has also been shown that PRFE triggers a genetic sequence or cascade of 'wound repair' genes critical for the four stages of wound healing: inflammation, granulation, epithelialization, and remodeling.
* It has been utilized in the VA Health System since 2004 with no serious adverse events attributable to the device.

This study will assess as an endpoints:

* Primary - the incidence of wounds reaching complete closure, and
* Secondary - the time to complete wound closure percentage reduction in wound area, percentage reduction in wound volume, and rate of healing mm2/day and mm3/day.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females > 18 years of age
2. History of Type 1 or 2 Diabetes Mellitus
3. A diabetic plantar foot wound, Wagner grade 1 or 2 (See Exclusion Criteria, number four (4).
4. The qualifying wound must have been present for ≥ 30 days; (the age of the wound will be recorded) based on patient history or documentation in the medical record.
5. Ankle Brachial Index (ABI) score ≥ 0.7 and ≤ 1.2 with present palpable posterior tibial pulse or dorsalis pedis pulse in index foot
6. Wound surface area ≥ 1.0 cm2 and ≤ 16.0 cm2
7. Female subjects of childbearing age will be expected to test negative after taking a serum pregnancy test. Additionally, they must be willing to use an adequate and reliable method of contraception for the study duration. Females who are postmenopausal must have been postmenopausal at least one year or twelve months.

Exclusion Criteria:

1. Glycosylated Hemoglobin (HbA1c) greater than 12 within 30 days of enrollment
2. Absent pedal Doppler signals in the foot with the index wound or the presence of significant peripheral artery disease ,
3. Concurrent treatment of the index wound with another advanced wound care device (i.e. negative pressure wound therapy, non-contact ultrasound, hyperbaric oxygen, electrical stimulation) or pharmaceutical (e.g. growth factors) within thirty (30) days of enrollment.
4. Index wounds with exposed muscle, ligament or tendon, or which probe to bone regardless of classification-See Inclusion Criteria no. two ( 2).
5. Wounds due to a nondiabetic etiology (e.g. venous stasis, arterial insufficiency, etc.)
6. Cellulitis, osteomyelitis, or other clinical evidence of infection involving the index wound.
7. History of malignancy
8. Concurrent use of high dose immunosuppressant or cytotoxic drugs
9. Implanted pacemaker or defibrillator
10. Metallic implant involving the index foot or ankle
11. Implanted system with a metallic lead
12. Pregnant or lactating females
13. Concurrent participation in another clinical trial. 14) An unwillingness of the patient to comply with the study procedures and the required follow-up regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Wilson, DPM, Principal Investigator — Winston - Salem Outpatient Clinic, WG Hefner VAMC
Locations (1):
- Winston - Salem Outpatient Clinic, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: standardized care will be used for wound care on patients randomized to this arm.
- Active: Provant Therapy Device
Period: Overall Study
Arm/Group | Standard of Care | Active
Started | 4 | 4
Completed | 2 | 3
Not Completed | 2 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active: The Provant Wound Therapy System: The Provant Wound Therapy System is a safe adjuvant non-invasive medical device.
- Standard of Care: Standardized wound care is used
- Total: Total of all reporting groups
Arm/Group | Active | Standard of Care | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Wounds Reaching Complete Closure
Time Frame: approximate one year
Population: Analysis was not done as this study was early terminated due to all subjects not meeting inclusion/exclusion criteria.
Groups:
- Active Provant Device: Active Device
  The Provant Wound Therapy System: The Provant Wound Therapy System is a safe adjuvant non-invasive medical device.
Arm/Group | Standard of Care | Active Provant Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard of Care | Active
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=4) | Active (N=4)
Death (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No